CLINICAL TRIAL: NCT03366571
Title: Improvement of Hard Endpoint in Chronic Hepatitis B Patients Treated With Antiviral Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking University First Hospital (Other); Peking University People's Hospital (Other); Beijing YouAn Hospital (Other); Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Jidong Jia, Director of Liver Research Center, Beijing Friendship Hospital
Other Study IDs: D161100002716003
Record Dates: First submitted 2016-07-29; First posted 2017-12-08 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Chronic Hepatitis B
Keywords: Liver Cirrhosis
MeSH Terms: conditions — Hepatitis B, Chronic; Liver Cirrhosis | interventions — entecavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma and DNA.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Anti-viral therapy group: Subjects who have completed the 3 years research "Clinical Effects and Cost-effectiveness Analysis of Early Anti-viral Therapy on HBV-related Compensated Liver Cirrhosis"
  Interventions: Drug: Nucleos(t)ide Analogues
- Non anti-viral therapy group: History study from literature

INTERVENTIONS:
Drug: Nucleos(t)ide Analogues — Entecavir 0.5mg daily, Lamivudine100mg qd daily, Adefovir Dipivoxil 10mg daily, telbivudine 600mg qd daily, their combination therapy, tenofovir 300mg qd daily.
  Other Names: Baraclude , et al
  Groups: Anti-viral therapy group

SUMMARY:
Patients who have completed 3 years follow-up of the past Beijing Science and Technology Commission Research will receive another 7-years anti-viral therapy. Patients will be assessed at baseline and every six months for blood cell count, liver function test, HBVDNA, AFP, prothrombin time, liver ultrasonography, and Fibroscan. CT or MRI and endoscopy will be performed at baseline and 7 years. At the end of the study, the cumulative rate of clinical hepatic hard endpoint will be calculated.

DETAILED DESCRIPTION:
Patients who have completed 3 years follow-up of the past Beijing Science and Technology Commission Research will receive another 7-years anti-viral therapy. Patients will be assessed at baseline and every six months for blood cell count, liver function test, HBVDNA, AFP, prothrombin time, liver ultrasonography, and Fibroscan. CT or MRI and endoscopy will be performed at baseline and 7 years. At the end of the study, the cumulative rate of clinical hepatic hard endpoint will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have participated in the research funded by Beijing science and Technology Commission and have completed 156 weeks follow-up.
* Patients comply with the requirements of the trail voluntarily
* Written informed consent

Exclusion Criteria:

* Pregnant woman or patient with severe disease
* Patients with poor adherence to the study
* Patients not suitable for the study evaluated by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The HBV-related chronic hepatitis /cirrhosis patients who have completed 3 years follow-up of the past Beijing Science and Technology Commission Research.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-01; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative rate of liver decompensation and/or hepatic carcinoma and/or liver related death | 10 years
  Cumulative rate of liver decompensation (including ascites,hepatic encephalopathy,Gastrointestinal hemorrhage)，and/or hepatocellular carcinoma， and/or liver related death after 10 years of antiviral treatment

SECONDARY OUTCOMES:
HBV-DNA undetectable rate | 10 years
  HBV-DNA undetectable rate after 10 years of antiviral treatment
Decrease of transient elastography | 10 years
  Decrease of transient elastography after 10 years of antiviral treatment
HBeAg seroconversion rate | 10 years
  HBeAg seroconversion rate after 10 years of antiviral treatment
HBsAg seroconversion rate | 10 years
  HBsAg seroconversion rate after 10 years of antiviral treatment
Decrease of Child-Pugh score | 10 years
  Decrease of Child-Pugh score after 10 years of antiviral treatment
Decrease of MELD score | 10 years
  Decrease of MELD score after 10 years of antiviral treatment
Improvement of life Quality assessed by SF-36 | 10 years
  Improvement of life Quality assessed by SF-36 after 10 years of antiviral treatment
Improvement of life Quality assessed by EQ-5D | 10 years
  Improvement of life Quality assessed by EQ-5D after 10 years of antiviral treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dong J Jia, Doctor, Principal Investigator — Beijing Friendship Hospital
Locations (4):
- China (4):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Beijing, Beijing Municipality
  - Peking University People's Hopsital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wu X, Zhou J, Sun Y, Ding H, Chen G, Xie W, Piao H, Xu X, Jiang W, Ma H, Ma A, Chen Y, Xu M, Cheng J, Xu Y, Meng T, Wang B, Chen S, Shi Y, Kong Y, Ou X, You H, Jia J. Prediction of liver-related events in patients with compensated HBV-induced cirrhosis receiving antiviral therapy. Hepatol Int. 2021 Feb;15(1):82-92. doi: 10.1007/s12072-020-10114-1. Epub 2021 Jan 18. PMID 33460002